CLINICAL TRIAL: NCT03194412
Title: FOCUS- Frailty Management Optimization Through EIP AHA Commitments and Utilization of Stakeholders Input (WP7-WMU)
Brief Title: FOCUS- Frailty Management Optimization Through EIP AHA Commitments and Utilization of Stakeholders Input
Acronym: FOCUS-WMU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wroclaw Medical University (Other)
Collaborators: University of Valencia (Other); Roessingh Research and Development (Other); Aston Research Centre for Healthy Ageing (ARCHA) (Unknown); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); Nursing School of Coimbra (ESEnfC) (Unknown); Aveiro University (Other); EVERIS (Unknown); Advanced Software Studies And Maintenance Of Technology (Other)
Responsible Party: Principal Investigator, Donata Kurpas, Donata Kurpas, MD, PhD, Assoc. Prof., Wroclaw Medical University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 664367/FOCUS; 664367/FOCUS (Other Grant/Funding Number: EU HP and Ministry of Science and Higher Education in Poland)
Record Dates: First submitted 2017-06-17; First posted 2017-06-21 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Frailty
Keywords: Frail Elderly; Geriatric Assessment; Humans; Aged
MeSH Terms: conditions — Frailty | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: The group of participants involved to the study:
  * n=60 ( at least 30) to diet /nutritional - intervention group 1
  * n=60 ( at least 30) to physical activity - intervention group 2
  * n=60 ( at least 30) to comprehensive therapy (diet/nutritional+physical activity training) - intervention group 3
  * n=30 (at least 15) formal and informal caregivers of elderly - intervention group 4
  * n=60 ( at least 30) to control group without intervention - group 5
  Evaluation process:
  * Screening Evaluation (stage 1)- investigated within 0
  * Baseline Evaluation (stage 2) - after 3 months from 0
  * Final Evaluation (stage 3) - after 6 months from 0 Professionals involved in the interventions: physicians, general practitioners, physiotherapists, rehabilitation professionals, educators, nurses, volunteers, nutrition consultant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Diet /nutritional (Experimental): Special diet for elderly. It should be rich in the appropriately amount of protein, carotenoids, vitamins, minerals, macro and micronutrients.
  Interventions: Dietary Supplement: Diet /nutritional
- Physical activity (Experimental): Regular physical activity in everyday life of the elderly - exercises to improve coordination and balance, stretching exercises, strength exercises.
  Interventions: Behavioral: Physical activity
- Comprehensive therapy (Experimental): Special diet for elderly (appropriately amount of protein, carotenoids, vitamins, minerals, macro and micronutrients) and regular physical activity in everyday life of the elderly (exercises to improve coordination and balance, stretching exercises, strength exercises)
  Interventions: Combination Product: Comprehensive therapy
- Caregivers of elderly (Experimental): Education about frailty: prevention and treatment (nutrition, physical activity, dietary supplement diet).
  Interventions: Behavioral: Caregivers of elderly
- Control group (No Intervention): Without intervention

INTERVENTIONS:
Dietary Supplement: Diet /nutritional — • Duration:
  * the first stage - 3 months: 12 weeks
  * second stage - 3 months: 12 weeks
  Each patient collect a detailed menu of the last two days before making the description. Then the menu is analyzed by a nutrition consultant. The role of nutrition consultant is:
  * make a diet modification to include the products recommended in frailty
  * modifying eating habits
  The diet modification is mainly focused on adequate supply:
  * vitamin D (according to Central Europe guidelines -2013 for seniors)
  * protein (according to European Society for Clinical Nutrition and Metabolism (ESPEN recommendations)
  Arms: Diet /nutritional
Behavioral: Physical activity — * Duration:
    * the first stage - 3 months: 12 weeks
    * second stage - 3 months: 12 weeks
  * Frequency: twice a week
  * Duration of each session: 60 minutes
  Worksheets for the elderly with frailty syndrome have been developed:
  * resistance exercises and strength training, which aim to improve muscle strength in the limbs
  * exercises aimed at improving motor coordination, flexibility and speed
  * stretching exercises.
  Other Names: regular physical activity in everyday life of the elderly
  Arms: Physical activity
Combination Product: Comprehensive therapy — Combination of special diet for elderly (as in Group 1) and regular physical activity into everyday life of the elderly (as in Group 2)
  Duration:
  * the first stage - 3 months- 12 weeks
  * the second stage - 3 months- 12 weeks Frequency of physical activity: twice a week Duration of each session: 60 minutes
  Other Names: diet/nutritional and physical activity training
  Arms: Comprehensive therapy
Behavioral: Caregivers of elderly — Group: formal and informal caregivers of elderly with frailty syndrome Materials and Tools: multimedia presentation about frailty prevention and treatment (nutrition, physical activity, dietary supplement diet).
  Duration:
  * the first stage - 3 months: 12 weeks
  * the second stage - 3 months: 12 weeks
  Frequency: 1 (at the beginning of stage 0, 1 and 2) Duration: 60 minutes
  Arms: Caregivers of elderly

SUMMARY:
This intervention study is a part of the FOCUS (Frailty Management Optimization Through EIP AHA Commitments and Utilization of Stakeholders Input) project which purpose is to critically reduce the burden of frailty in Europe by assisting those partners within the European Innovation Partnership for Active Healthy Ageing (EIPAHA) with commitments focusing on early diagnosis/ screening and/or management of frailty to achieve scalability.

FOCUS aims to critically reduce the burden of frailty in Europe by developing methodologies and tools to assist entities focusing on early diagnosis, screening and management of frailty to achieve scalability. Frailty is a common clinical syndrome in older adults that brings an increased risk for poor health outcomes including falls, incident disability, hospitalization and mortality.

The FOCUS Consortium brings together a multidisciplinary team of specialists from 10 organizations in 6 countries - Italy, Poland, Portugal, Spain, Netherlands, United Kingdom - that will work on developing, piloting and disseminating methodologies and tools to assist entities focusing on early diagnosis, screening and management of frailty to achieve scalability.

Wroclaw Medical University actively participates in all projects for the advances in science, entrepreneurship, technological innovation, both with public authorities, local governments, and enterprises. In FOCUS project, WMU is responsible for Evaluation of the project and collaborates with the others partners in Coordination of the project, Dissemination of the project, Synthesis of learning and realities of practice, Analysis and guidelines development, Creation of Network and Platform for knowledge exchange, Test of guidelines in a set of commitments (Work Package 7 - WP7).

The outcomes of this proposal will offer significant potential improvements for innovative, coordinated and comprehensive community based prevention with regard to the optimisation of functional capacity tools to address pre-frailty, and for improving the management of frailty.

The registered study has its own protocol developed by Wroclaw Medical University research team and will be implemented within WP7 of the FOCUS project.

DETAILED DESCRIPTION:
This is a prospective intervention study. The study is expected screening about 320 participants - persons aged more than 60 years old recruited from Universities of the Third Age, day care centers, primary care centers, geriatrics out-patient clinics and from nursing homes. We are expected to enroll 270 potential participants (at least 135 participants) to 5 groups: 4 intervention groups and 1 control group without any intervention.

Patient qualification is based on criteria developed by Fried et al 2001.

Dimensions:

Weight loss Exhaustion Physical Activity Walk Time Grip Strength

INTERPRETATION:

Robust: 0 points Pre-frail: 1-2 points Frail: 3 or more points

Method: diagnostic survey Technique: the 'surveys combined with direct measurements of patients investigated within 0, after 3 and 6 months

Tools:

Study questionnaires:

• Standardized questionnaires: Center for Epidemiologic Studies Depression Scale Minnesota Leisure Time Physical Activity Questionnaire Vulnerable Elders - 13 Survey Mini Nutritional Assessment Health Behaviour Inventory Montreal Cognitive Assessment Geriatric Depression Scale World Health Organization Quality of Life (short version) questionnaire Camberwell Assessment of Need Short Appraisal Schedule Barthel Scale Activities of Daily Living Instrumental Activities of Daily Living Camberwell Assessment of Need Short Appraisal Schedule Timed up and go test Beck Depression Inventory

* The questionnaire on: socio-demographic data - age, gender, marital status, living in relationship/ without relationship, level of education, place of residence, economic status; the number of hospitalizations in the last 3 years (including kind of ward); the number and kind of chronic diseases (ICD-10); the number of permanent medications; employment situation; number of traveling in the last year; having pets; number of languages the participants can speak; number of falls
* Rating of patients' difficulties in the implementation of the intervention (Did the patients perform the interventions? How often? Was it difficult to the patients?)
* Observations sheet: height, weight, BMI, hand grip strength, circumference of arm muscle, circumference of calf
* The results of laboratory tests: sodium , albumins, lymphocytes, LDL cholesterol, C reactive proteins, glomerular filtration rate, fasting glucose, thyroid hormones

ELIGIBILITY:
Inclusion Criteria:

* patients:

  * age ≥ 60 years old
  * recognition of the pre-frail and frail (based on the scale of the Cardiovascular Health Study)
  * consent to participate in the study
  * the patients who could speaking Polish language
* caregivers:

  * to be formal or informal caregivers of person aged ≥ 60 years old
  * consent to participate in the study
  * caregivers who could speaking Polish language

Exclusion Criteria:

* patients:

  * age < 60 years old
  * lack of recognition of the pre-frail and frail (based on the scale of the Cardiovascular Health Study)
  * somatic state which precludes complete examination performance according to selected scales (eg. Vision disorders)
  * severe mental disorders or difficulties that prevent active participation in the study
  * the patients who could not speaking Polish language
  * lack of consent to participate in the study
* caregivers:

  * not to be formal or informal caregivers of person aged ≥ 60 years old
  * lack of consent to participate in the study
  * the caregivers who could not speaking Polish language

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Functional status change | 6 months
  People who improved/worsened functional status according to standardized measures

SECONDARY OUTCOMES:
Falls change | 6 months
  People who had at least one fall during the period of the intervention
Mood change | 6 months
  People who improved/worsened mood status according to standardized measures
Nutritional status change | 6 months
  People who improved /worsened nutritional status according to standardized measures
Cognitive status change | 6 months
  People who improved /worsened cognitive status according to standardized measures

CONTACTS AND LOCATIONS:
Overall Officials: Aneta Soll, MSc, Principal Investigator — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonio Cano, Donata Kurpas, Maria Magdalena Bujnowska-Fedak, Silvina Santana, Carol Holland, Maura Marcucci, Ana Gonzalez- Segura, Miriam Vollenbroek-Hutten, Barbara D'Avanzo, Alessandro Nobili, João Luís Al ves Apostolo, Elżbieta Bobrowicz-Campos, Ana M. Martínez-Arroyo. FOCUS: Frailty Management Optimisation through EIPAHA Commitments and Utilisation of Stakeholders' Input - an innovative European Project in elderly care. Family Medicine & Primary Care Review 2016; 18, 3: 373-376 DOI: https://doi.org/10.5114/fmpcr/63234
- [Background] Piotrowicz J, Soll A, Kielar U, Zwiefka A, Guligowska A, Pigłowska M, Kostka T, Kurpas D. ICT and environmental support for patients with frailty syndrome: CareWell Project, Focus Project and SUNFRAIL Project. Medical Science Pulse 2017; 11, 1: 37-43.
- See also: Family Medicine & Primary Care Review — https://www.termedia.pl/FOCUS-Frailty-Management-Optimisation-through-EIPAHA-Commitments-and-Utilisation-of-Stakeholders-Input-an-innovative-European-Project-in-elderly-care-,95,28467,0,1.html
- See also: Medical Science Pulse — http://medicalsciencepulse.com/resources/html/article/details?id=146026